CLINICAL TRIAL: NCT06010030
Title: A Randomized Clinical Trial of TDCS to Remediate Phonological Impairment in Aphasia
Brief Title: HD-tDCS for Phonological Impairment in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Priyanka Shah-Basak, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00046308
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Intervention Model Description: Participants will maintain one of two speech therapy modalities throughout the study and be assigned to either targeted anodal-tDCS or sham-tDCS.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Care provider, participant, and outcome assessor are masked for tDCS status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HD-tDCS (Experimental): Participants will be randomized to receive either anodal HD-tDCS or sham-tDCS.
  Interventions: Device: Targeted Transcranial Direct Current Stimulation
- Speech Therapy (Experimental): Participants will be randomized to receive either phonologic-focused speech therapy or semantic-focused speech therapy
  Interventions: Behavioral: Speech Therapy

INTERVENTIONS:
Device: Targeted Transcranial Direct Current Stimulation — High-Definition-tDCS will be delivered via a battery-driven constant direct current stimulator (Soterix) using a 4x1 montage (1 central anodal electrode and 4 cathodal electrodes) arranged in a HD-cap. Anodal or sham tDCS will be administered.
  Other Names: HD-tDCS; tDCS
  Arms: HD-tDCS
Behavioral: Speech Therapy — Participants will receive either semantic or phonological focused speech therapy
  Arms: Speech Therapy

SUMMARY:
This study will investigate the effects of mild electrical stimulation in conjunction with speech therapy for people with post-stroke aphasia to enhance language recovery.

DETAILED DESCRIPTION:
Aphasia is a disturbance of language, primarily caused by brain injury to the left cerebral hemisphere. Aphasia treatments include speech and language therapy and pharmacologic therapy, but several studies have found that these treatments are not completely effective for patients with aphasia, leaving them with residual deficits that significantly add to the cost of stroke-related care. Additionally, the amount and frequency of speech and language therapy delivered may have a critical effect on recovery. Therefore, there is a need for new treatments or adjuncts to existing treatments, such as brain stimulation interventions, that have the potential to show greater improvements in patients with aphasia. One such new approach for non-invasive brain stimulation is transcranial direct current stimulation (tDCS).

This study will examine the effects of tDCS during speech therapy to further examine which method or methods is best for patient recovery. Patients enrolled in the study will undergo language testing that covers a broad range of language functions. Functional Magnetic Resonance Imaging (fMRI) will be completed before and after speech therapy intervention arms to investigate the neural processes affected by tDCS and speech therapy.

Study design:

Patients will be randomly assigned to one of 2 speech therapy groups as well as randomly assigned to one of 2 stimulation groups (active anodal stimulation or sham). Patients will receive one of two different speech therapy treatment interventions to focus on specific processing deficits. Participants will undergo neuropsychological evaluation and fMRI assessment before receiving targeted anodal-tDCS or sham-tDCS for 10 therapy sessions. Participants will then be re-tested using the behavioral assessment measure and fMRI before crossing over to receive the tDCS intervention again, along with the same speech therapy arm. They will complete a behavioral assessment and fMRI at 3 months post Treatment 2 and a final behavioral assessment at 6 months post Treatment 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 or older.

Patients may not be older than 85.

Patients must have a language deficit from left-sided focal neurologic damage (e.g. stroke, tumor).

Patients must be adults and have English-language fluency.

Patients must be eligible to undergo MRI.

Beyond meeting the inclusion criteria, no preference will be given on the basis of race, ethnicity or gender.

Exclusion Criteria:

* Advanced neurodegenerative disease (i.e. Stage 3 Alzheimer's disease)

Neurologic disease (e.g. idiopathic epilepsy, seizure disorders that are not well managed, Parkinson's disease, ALS),

Severe psychopathology (e.g. schizophrenia, bipolar disorder, acute major depressive episode)

Suspected or diagnosed uncorrectable hearing or vision difficulties, or developmental disabilities (i.e. intellectual disability or learning disability).

Contraindications to MRI such as claustrophobia, implanted electronic devices, MRI-incompatible metal in the body, extreme obesity, pregnancy, inability to lie flat, inability to see or hear stimulus materials.

Younger than 18 or older than 85.

< 6 months post tumor resection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral outcome | Upon the completion of therapy cycle (a cycle consists of 10 intervention days) and 10 weeks post completion of therapy
  Percent improvement on behavioral outcomes after each therapy cycle will be the primary behavioral outcome measure.

SECONDARY OUTCOMES:
fMRI | 3 time points: pre-assessment, 10 weeks post-therapy cycle A and 10 weeks post-therapy cycle B
  fMRI functional changes between time points

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen PM, Vinter K, Olsen TS. Aphasia after stroke: type, severity and prognosis. The Copenhagen aphasia study. Cerebrovasc Dis. 2004;17(1):35-43. doi: 10.1159/000073896. Epub 2003 Oct 3. PMID 14530636
- [Background] Greener J, Enderby P, Whurr R. Pharmacological treatment for aphasia following stroke. Cochrane Database Syst Rev. 2001;2001(4):CD000424. doi: 10.1002/14651858.CD000424. PMID 11687079
- [Background] Kelly H, Brady MC, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2010 May 12;(5):CD000425. doi: 10.1002/14651858.CD000425.pub2. PMID 20464716
- [Background] Lincoln NB, McGuirk E, Mulley GP, Lendrem W, Jones AC, Mitchell JR. Effectiveness of speech therapy for aphasic stroke patients. A randomised controlled trial. Lancet. 1984 Jun 2;1(8388):1197-200. doi: 10.1016/s0140-6736(84)91690-8. PMID 6202993
- [Background] Ellis C, Simpson AN, Bonilha H, Mauldin PD, Simpson KN. The one-year attributable cost of poststroke aphasia. Stroke. 2012 May;43(5):1429-31. doi: 10.1161/STROKEAHA.111.647339. Epub 2012 Feb 16. PMID 22343643
- [Background] Ellis C, Dismuke C, Edwards KK. Longitudinal trends in aphasia in the United States. NeuroRehabilitation. 2010;27(4):327-33. doi: 10.3233/NRE-2010-0616. PMID 21160122
- [Background] Boysen AE, Wertz RT. Clinician Costs in Aphasia Treatment: How Much Is a Word Worth? Clin. Aphasiology 1996;24:207-213
- [Background] Meinzer M, Djundja D, Barthel G, Elbert T, Rockstroh B. Long-term stability of improved language functions in chronic aphasia after constraint-induced aphasia therapy. Stroke. 2005 Jul;36(7):1462-6. doi: 10.1161/01.STR.0000169941.29831.2a. Epub 2005 Jun 9. PMID 15947279
- [Background] Holland R, Crinion J. Can tDCS enhance treatment of aphasia after stroke? Aphasiology. 2012 Sep;26(9):1169-1191. doi: 10.1080/02687038.2011.616925. Epub 2011 Nov 3. PMID 23060684
- [Background] Paulus W. Transcranial direct current stimulation (tDCS). Suppl Clin Neurophysiol. 2003;56:249-54. doi: 10.1016/s1567-424x(09)70229-6. PMID 14677402
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. Brain. 2002 Oct;125(Pt 10):2238-47. doi: 10.1093/brain/awf238. PMID 12244081
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Darkow R, Martin A, Wurtz A, Floel A, Meinzer M. Transcranial direct current stimulation effects on neural processing in post-stroke aphasia. Hum Brain Mapp. 2017 Mar;38(3):1518-1531. doi: 10.1002/hbm.23469. Epub 2016 Nov 11. PMID 27859982
- [Background] Meinzer M, Jahnigen S, Copland DA, Darkow R, Grittner U, Avirame K, Rodriguez AD, Lindenberg R, Floel A. Transcranial direct current stimulation over multiple days improves learning and maintenance of a novel vocabulary. Cortex. 2014 Jan;50:137-47. doi: 10.1016/j.cortex.2013.07.013. Epub 2013 Aug 6. PMID 23988131
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Cohen Kadosh R, Soskic S, Iuculano T, Kanai R, Walsh V. Modulating neuronal activity produces specific and long-lasting changes in numerical competence. Curr Biol. 2010 Nov 23;20(22):2016-20. doi: 10.1016/j.cub.2010.10.007. Epub 2010 Nov 4. PMID 21055945
- [Background] Vestito L, Rosellini S, Mantero M, Bandini F. Long-term effects of transcranial direct-current stimulation in chronic post-stroke aphasia: a pilot study. Front Hum Neurosci. 2014 Oct 14;8:785. doi: 10.3389/fnhum.2014.00785. eCollection 2014. PMID 25352798
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Pillay SB, Stengel BC, Humphries C, Book DS, Binder JR. Cerebral localization of impaired phonological retrieval during rhyme judgment. Ann Neurol. 2014 Nov;76(5):738-46. doi: 10.1002/ana.24266. Epub 2014 Sep 19. PMID 25164766
- [Background] Saffran EM, Marin OS. Reading without phonology: evidence from aphasia. Q J Exp Psychol. 1977 Aug;29(3):515-25. doi: 10.1080/14640747708400627. No abstract available. PMID 905501
- [Background] Caramazza A, Berndt RS, Basili AG. The selective impairment of phonological processing: a case study. Brain Lang. 1983 Jan;18(1):128-74. doi: 10.1016/0093-934x(83)90011-1. PMID 6839129
- [Background] Kohn SE. Conduction Aphasia. Psychology Press; 2013.
- [Background] Pillay SB, Gross WL, Graves WW, Humphries C, Book DS, Binder JR. The Neural Basis of Successful Word Reading in Aphasia. J Cogn Neurosci. 2018 Apr;30(4):514-525. doi: 10.1162/jocn_a_01214. Epub 2017 Dec 6. PMID 29211656
- [Background] Binder JR, Desai RH, Graves WW, Conant LL. Where is the semantic system? A critical review and meta-analysis of 120 functional neuroimaging studies. Cereb Cortex. 2009 Dec;19(12):2767-96. doi: 10.1093/cercor/bhp055. Epub 2009 Mar 27. PMID 19329570
- [Background] U.S. Census Bureau. State & County QuickFacts: Milwaukee County, Wisconsin [Internet]. [date unknown];[cited 2018 Jan 11 ] Available from: https://factfinder.census.gov/faces/tableservices/jsf/pages/productview.xhtml?src=CF
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Wilson SM, Yen M, Eriksson DK. An adaptive semantic matching paradigm for reliable and valid language mapping in individuals with aphasia. Hum Brain Mapp. 2018 Aug;39(8):3285-3307. doi: 10.1002/hbm.24077. Epub 2018 Apr 17. PMID 29665223
- [Background] Yen M, DeMarco AT, Wilson SM. Adaptive paradigms for mapping phonological regions in individual participants. Neuroimage. 2019 Apr 1;189:368-379. doi: 10.1016/j.neuroimage.2019.01.040. Epub 2019 Jan 18. PMID 30665008
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622